CLINICAL TRIAL: NCT00354874
Title: A Multi-centre, Randomised, Double-blind, Placebo Controlled, Dose Ascending, Four Way Crossover Study to Examine Efficacy (FEV1), Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Single and Repeat Doses of GW642444
Brief Title: Investigation Of A New Medication (GW642444) In Asthmatic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B2C101762
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: GW642444 asthmatic subjects safety tolerability PD and PK
MeSH Terms: conditions — Asthma | interventions — Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- GW642444 50mcg (Experimental)
  Interventions: Drug: GW642444
- GW642444 100mcg (Experimental)
  Interventions: Drug: GW642444
- GW642444 200mcg (Experimental)
  Interventions: Drug: GW642444
- salmeterol 50mcg (Active Comparator)
  Interventions: Drug: salmeterol 50mcg
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GW642444 — drug
  Arms: GW642444 100mcg; GW642444 200mcg; GW642444 50mcg
Drug: Placebo — placebo
  Arms: placebo
Drug: salmeterol 50mcg — salmeterol
  Arms: salmeterol 50mcg

SUMMARY:
This study will evaluate efficacy (FEV1), safety, tolerability, pharmacodynamics and pharmacokinetics of single and repeat inhaled doses of GW642444. This will be a multi-centre, double-blind, placebo controlled, dose ascending, four way cross-over study in approximately 28 mild to moderate asthmatic subjects.

Key assessments: Efficacy, safety, tolerability, pharmacodynamics and pharmacokinetics will be assessed by measurement of FEV1, blood pressure, heart rate, 12-lead ECGs, clinical laboratory tests, collection of adverse events (AE) information and blood samples.

ELIGIBILITY:
Inclusion criteria:

* Female subjects must be non-childbearing (i.e., surgically sterilised or post-menopausal).
* Non-smokers for at least 6 months.
* Stable asthma.

Exclusion criteria:

* Abnormal findings on heart monitoring assessment.
* Lower respiratory tract infection within 4 weeks, upper respiratory tract within 2 weeks of study.
* Currently taking doses of fluticasone propionate over 500mcg/day.
* Unstable asthma medication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-01; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
FEV1 at 24 hours after a single dose. | 24 hours on 4 separate occasions

SECONDARY OUTCOMES:
FEV1 - Days 1 and 7 | Days 1 and 7 on 4 separate occasions
Mean morning/evening PEFR | Days 3-8 on 4 separate occasions
BP, HR & QTc on Days 1 and 7 | Days 1 and 7 on 4 separate occasions
Potassium and glucose on Days 1 and 7 | Days 1 and 7 on 4 separate occasions
safety & tolerability as measured by AEs, laboratory safety tests, cardiac monitoring, VS & ECG | throughout study
PK parameters | Days 1, 4 and 7 on 4 separate occasions

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Germany (2):
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
- GSK Investigational Site, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: B2C101762 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: B2C101762 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: B2C101762 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: B2C101762 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: B2C101762 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: B2C101762 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: B2C101762 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register